CLINICAL TRIAL: NCT04563546
Title: Community and Physician Perceptions of Chest Pain and Prevalence of Acute Coronary Syndrome Among HIV-infected and -Uninfected Patients in Moshi, Tanzania
Brief Title: Acute Coronary Syndrome KCMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00090902
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MI Patients in northern Tanzania (Other): Patients presenting to KCMC emergency department with acute MI
  Interventions: Other: Quality Improvement

INTERVENTIONS:
Other: Quality Improvement — A quality improvement intervention including reminders, care protocols, and text messages to improve care of myocardial infarction in the KCMC ED

SUMMARY:
The purpose of this study is to develop a quality improvement intervention to address barriers to evidence-based acute coronary syndrome (ACS) care in northern Tanzania. Patients who presented to Kilimanjaro Christian Medical Center (KCMC) will be asked to complete a survey about barriers and facilitators of health care. In addition the survey will be administered to all providers, policymakers, and administrators participating in in-depth interviews. Data from this survey will be used to develop a quality improvement intervention that will be piloted by KCMC staff. Six months after the pilot program is implemented providers, patients, and administrators will be interviewed for their perspectives on the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* symptoms related to acute coronary syndrome
* myocardial infarction
* clinically sober
* able to communicate in Swahili or English

Exclusion Criteria:

* medically unstable
* have a deteriorating condiction
* too critically ill to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Hertz, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We are bound by local Tanzanian guidelines regarding patient privacy and data security and are not allowed to share individual participant data without express permission of the Tanzanian National Institute for Medical Research.

REFERENCES:
- [Derived] Hertz JT, Nworie JE, Shayo F, Galson SW, Coaxum LA, Daniel I, Makambay PS, Akrabi AM, Manyangu GJ, Thielman NM, Bloomfield G, Sakita FM. Acute myocardial infarction diagnosis and treatment following implementation of a multicomponent intervention in Tanzania: the MIMIC pilot trial. BMJ Open. 2025 Nov 11;15(11):e107857. doi: 10.1136/bmjopen-2025-107857. PMID 41218933
- [Derived] Hertz JT, Sakita FM, Haukila KF, Shayo PS, Shayo FM, Willy J, Lameck G, Kisanga E, Bosworth HB, Bettger JP, Rahim FO. Acceptability and Feasibility of a Multicomponent Intervention to Improve Acute Myocardial Infarction Care in Northern Tanzania: the MIMIC Pilot Trial. medRxiv [Preprint]. 2024 Dec 16:2024.12.13.24319026. doi: 10.1101/2024.12.13.24319026. PMID 39763513
- [Derived] Hertz JT, Sakita FM, Rahim FO, Mmbaga BT, Shayo F, Kaboigora V, Mtui J, Bloomfield GS, Bosworth HB, Bettger JP, Thielman NM. Multicomponent Intervention to Improve Acute Myocardial Infarction Care in Tanzania: Protocol for a Pilot Implementation Trial. JMIR Res Protoc. 2024 Sep 24;13:e59917. doi: 10.2196/59917. PMID 39316783

RESULTS

PARTICIPANT FLOW:
Groups:
- Myocardial Infarction (MI) Patients in Northern Tanzania: Patients presenting to KCMC (Kilimanjaro Christian Medical Center) emergency department with acute MI
  Quality Improvement: A quality improvement intervention including reminders, care protocols, and text messages to improve care of myocardial infarction in the KCMC ED
- Providers in the KCMC Emergency Department: Providers in the KCMC (Kilimanjaro Christian Medical Center) Emergency Department
Period: Overall Study
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania | Providers in the KCMC Emergency Department
Started | 577 | 64
Completed | 577 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania | Providers in the KCMC Emergency Department | Total
Number analyzed (Participants) | 577 | 64 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (18.0) | 29.6 (5.7) | 59.1 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 23 | 327
  Male | 273 | 41 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 577 | 64 | 641
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 577 | 64 | 641
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 577 | 64 | 641

OUTCOME MEASURES:

1. Primary Outcome: Acceptability as Measured by the Acceptability of Intervention Measure (AIM)
Description: The AIM tool is a 4-question survey that evaluates the acceptability of an intervention. Responses to each question are on a 5-point Likert Scale (Strongly Agree=5, Agree=4, Neutral=3, Disagree=2, Strongly Disagree=1). Responses of "Strongly Agree" (5) and "Agree" (4) are considered to indicate a more acceptable intervention. The responses to each question will be averaged together to give an acceptability score between 1 and 5 for each respondent. The primary outcome will be the overall mean acceptability score among respondents. A mean acceptability score >= 4 will be considered to indicate acceptability.
Time Frame: Initial ED visit (baseline)
Population: The AIM was assessed among KCMC ED providers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers in the KCMC Emergency Department
Number analyzed (Participants) | 64
score on a scale | 4.82 (0.31)

2. Secondary Outcome: Number of Participants Presenting With Chest Pain or Shortness of Breath Who Undergo ECG and Cardiac Biomarker Testing During Their ED Stay
Time Frame: Initial ED visit (baseline)
Measure: Count of Participants; unit: Participants
Groups:
- Myocardial Infarction (MI) Patients in Northern Tanzania: Patients presenting to KCMC emergency department with acute MI
  Quality Improvement: A quality improvement intervention including reminders, care protocols, and text messages to improve care of myocardial infarction in the KCMC ED
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania
Number analyzed (Participants) | 577
Participants | 431
Statistical Analysis 1: Comparison: Myocardial Infarction (MI) Patients in Northern Tanzania; Test type: Other; p < 0.001, Chi-squared — Unadjusted p-value. Threshold for statistical significance = 0.05

3. Secondary Outcome: Survival of Participants With Acute Coronary Syndrome (ACS) at 30 Days After Enrollment
Description: Number of participants with ACS who have survived at 30 days
Time Frame: 30 days after enrollment
Population: Participants who met criteria for ACS.
Measure: Count of Participants; unit: Participants
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania
Number analyzed (Participants) | 141
Participants | 90
Statistical Analysis 1: Comparison: Myocardial Infarction (MI) Patients in Northern Tanzania; Test type: Other; p = 0.739, Chi-squared

4. Secondary Outcome: Number of Participants With Acute Coronary Syndrome (ACS) Taking Aspirin at Baseline
Time Frame: Initial ED visit (baseline)
Population: Participants who met criteria for ACS.
Measure: Count of Participants; unit: Participants
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania
Number analyzed (Participants) | 141
Participants | 101
Statistical Analysis 1: Comparison: Myocardial Infarction (MI) Patients in Northern Tanzania; Test type: Other; p < 0.001, Chi-squared — Unadjusted p-value. Threshold for statistical significance = 0.05

5. Secondary Outcome: Number of Participants With Acute Coronary Syndrome (ACS) Taking Aspirin 30 Days After Enrollment
Time Frame: 30 days after enrollment
Population: Participants who met criteria for ACS and survived to 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania
Number analyzed (Participants) | 90
Participants | 42

ADVERSE EVENTS:
Time Frame: 30 days
Description: Any Adverse Event plausibly due to the intervention was collected.
Arm/Group | Myocardial Infarction (MI) Patients in Northern Tanzania | Providers in the KCMC Emergency Department
All-Cause Mortality (participants affected / at risk) | 163/577 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/577 | 0/64
Other Adverse Events (participants affected / at risk) | 0/577 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT04563546/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04563546/ICF_000.pdf